CLINICAL TRIAL: NCT01909128
Title: Fermented Milk and Fermented Rice on the Appearance of Respiratory and Gastrointestinal Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 210/12
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Gastrointestinal Infections; Respiratory Infections
Keywords: children, fermented milk fermented rice, gastrointestinal infections, respiratory infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Cultured Milk Products

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- fermented milk (Experimental)
  Interventions: Dietary Supplement: fermented milk
- fermented rice (Experimental)
  Interventions: Dietary Supplement: fermented rice
- placebo (Placebo Comparator)

INTERVENTIONS:
Dietary Supplement: fermented milk — fermented milk with Lactobacillus CBA-L74
  Arms: fermented milk
Dietary Supplement: fermented rice — fermented rice wit Lactobacillus CBA-L74
  Arms: fermented rice

SUMMARY:
The respiratory and gastrointestinal infections are a very common problem with high morbidity in children. These conditions were due, in general, immaturity and all "inexperience" of the immune system, as well as to the particular anatomical structure and function of the respiratory and gastrointestinal tract still developing. This inevitably means that school-age children develop disease (as a result of infection) more easily than at later ages. The frequency and duration of these conditions implies a high discomfort and incur significant costs in relation to drug administration, the need for hospitalization, days of absence from school and work days lost by parents.

Recently probiotics, defined as "microorganisms that prove able, once ingested in adequate amounts, exert beneficial functions for the body "have been proposed for the treatment of treatment of respiratory and gastrointestinal infections of childhood but only in recent years have been conducted controlled clinical trials that have conclusively proven effectiveness. All probiotics induce an immune response, the characteristics of which are related to the strain or the mixture of bacteria used. Recent studies have demonstrated positive effects of probiotics on the respiratory system, and in particular on the prevention and reduction of the severity of respiratory infections, probably mediated by an increase of cells that secrete Immunoglobulin A in bronchial mucosa. It 'been shown that probiotics can be a sure way to reduce the risk of early acute otitis media and the use of antibiotics for recurrent respiratory infections during the first year of life. Similar results were seen in a study conducted on a population of 326 children aged between 3 and 5 years, who found a decrease in the incidence of antibiotic use by over 65% and a reduction of days of absence of more than 25% among children treated with a probiotic. Many of the studied effects of probiotics, understandably, refer to the digestive system. These effects relate to both conditions paraphysiological (constipation) and more specifically in situations of illness.

Most of the studies carried out in recent years has demonstrated the efficacy of specific probiotics in reducing the symptoms in the pediatric population affected by infectious gastroenteritis. Probiotics reduce the duration of infectious diarrhea by 0.7 days and reduce the frequency of diarrheal episodes in the first few hours.

The microbiota on the other hand participates in the function of the mucosal barrier against the adhesion of pathogenic bacteria, crucial time for the start of the infectious process.

When this barrier function is altered by chemical agents, by antigens or by stressors of different nature, may manifest intestinal disorders, sometimes due to the growth of bacteria pathogens. Numerous experimental data suggest that probiotics can contribute to the reinforcement of the activities of gut mucosal barrier, in particular aspects affecting the functionality of the intestinal epithelial cells or macrophages.

More recently it has been shown that daily intake for 3 months of preparation with probiotics reduce the incidence and severity of the most common respiratory infections and limits the number of days of absence school children during the winter season.

It's scientifically recognized as some probiotic effects can also be obtained with the use of inactivated bacteria or bacterial components isolated (eg bacterial DNA). It has been recently proposed a modified definition of probiotic products as "prepared bacterial cells or bacterial components that have a beneficial effect on the health and welfare of the host".

Among these products "probiotic-like" fall ingredients object of this study: food ingredients (rice flour and skim milk) fermented, or in which has been made to grow a probiotic (Lactobacillus CBA-L74) that has been inactivated at the end of the fermentation process through a heat treatment. The benefits are attributable to bacterial components that remain in the final product (for example, DNA, cell wall, etc.) and factors produced during the fermentation (short chain fatty acids, bacterial proteins, etc.).

The main effects of these bacterial components relate to the stimulation of the gastrointestinal tract associated lymphoid tissue (GALT), through interaction with the immune cells via Toll-like receptors.

In addition, some components, such as proteins and peptides, may have a Bifidogenic activity and are available in the literature some studies that have demonstrated the ability of infant formula, milk-based fermented to reduce the severity of episodes of infectious diarrhea in children.

With this data, the Commission of the European Society of Nutrition Gastroenterology, Hepatology and Pediatric Nutrition (ESPGHAN) has defined this type of products are not only safe but to determine a potential prebiotic effect and the reduction of the severity of episodes of infectious diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* children aged 12-48 months attending educational program (either at nursery or primary school)

Exclusion Criteria:

* concomitant chronic/congenital diseases and disabilities,
* active tuberculosis,
* congenital cardiac defects,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac diseases,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* chronic pulmonary diseases,
* malformation of the GI tract,
* history of allergy,
* severe wasting (less than 3 Standard deviations of weight-for-height z score),
* diarrhea on admission,
* antibiotic,
* pre/pro/symbiotic or immunostimulants use within 2 weeks before study start.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 405 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of fermented milk and rice administered daily for a total duration of 3 months on the appearance of common respiratory and gastrointestinal infections in schoolchildren aged between 12 and 48 months. | 3 months
  fermented milk and fermented rice on the appearance of respiratory and gastrointestinal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

REFERENCES:
- [Derived] Nocerino R, Paparo L, Terrin G, Pezzella V, Amoroso A, Cosenza L, Cecere G, De Marco G, Micillo M, Albano F, Nugnes R, Ferri P, Ciccarelli G, Giaccio G, Spadaro R, Maddalena Y, Berni Canani F, Berni Canani R. Cow's milk and rice fermented with Lactobacillus paracasei CBA L74 prevent infectious diseases in children: A randomized controlled trial. Clin Nutr. 2017 Feb;36(1):118-125. doi: 10.1016/j.clnu.2015.12.004. Epub 2015 Dec 17. PMID 26732025